CLINICAL TRIAL: NCT04869150
Title: Cigli Training and Research Hospital Organization
Brief Title: Does Myocardial Bridge Appear More Frequently and Diffusely on Radial Access Coronary Angiography
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Oktay Senoz, Principal Investigator, Izmir Bakircay University
Other Study IDs: 223-205
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Bridge of Coronary Artery
Keywords: myocardial bridge; radial access coronary angiography
MeSH Terms: conditions — Myocardial Bridging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- those with myocardial bridges
  Interventions: Procedure: radial access coronary angiography
- those without myocardial bridges

INTERVENTIONS:
Procedure: radial access coronary angiography — The right radial artery was cannulated with a 6-f radial sheath after local infiltration with 2% lidocaine.All patients received 5000 units of unfractionated heparin, 100 - 200 μg (depending on blood pressure) of nitroglycerin and 5 mg of diltiazem unless there was an absolute contraindication to diltiazem and anticoagulants.Coronary angiography was performed using the standard Judkins' technique via right radial access with a 5-f diagnostic catheter
  Groups: those with myocardial bridges

SUMMARY:
Although the incidence of myocardial bridge (MB) has been defined in different conventional coronary angiography (CCA) studies,the frequency of MB in radial access coronary angiography (RACA) is unknown.The aim of this study was to determine the incidence of MB in patients undergoing RACA.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing radial access coronary angiography
* Have myocardial bridge

Exclusion Criteria:

* A history of coronary artery bypass grafting (CABG)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective evaluation was made of the coronary angiographies of 2600 consecutive patients who underwent radial access coronary angiography between January 2018 and February 2020
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Does Myocardial Bridge Appear More Frequently and Diffusely on Radial Access Coronary Angiography? | 1 month
  the incidence of MB able to be detected on RACA was much higher than reported in previous CCA studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Cigli Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No